CLINICAL TRIAL: NCT02606942
Title: Prevalence of Chondromalacia Patella Among Adolescent Dancers - Correlation Between Symptoms and Sonography Findings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Head of the Department of Orthopedic Rehabilitaion, Sheba Medical Center
Other Study IDs: SHEBA-2079-15-SMC
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Chondromalacia; Cartilage Diseases
Keywords: chondromalacia patellae (CMP); patella
MeSH Terms: conditions — Cartilage Diseases; Chondromalacia Patellae; Patella Fracture | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dancers with knee injury: A cohort of dancers with reported knee injury. Questionnaires, physical exam, US of the knee
  Interventions: Other: Questionnaires, physical exam, US of the knee
- Dancers with no knee injury: A cohort of dancers without reported knee injury. Questionnaires, physical exam, US of the knee
  Interventions: Other: Questionnaires, physical exam, US of the knee
- Non-dancers athletes: A cohort of non-dancers athletes without knee injuries. Questionnaires, physical exam, US of the knee
  Interventions: Other: Questionnaires, physical exam, US of the knee

INTERVENTIONS:
Other: Questionnaires, physical exam, US of the knee — Function and pain questioners, physical findings and sonographic study of the knee joint

SUMMARY:
Comparing the physical and sonographic findings of dancers with Chondromalacia patella to non-dancers athletes.

DETAILED DESCRIPTION:
A cross sectional study in which comparing of dancers to non-dancers athletes will be carried. Specifically, chondromalacia patella will be studied and compared between dancers with and without knee injuries and non-dancers athletes.

Study will include detailed function and pain questionnaires, physical findings and sonographic study of the knee joint.

ELIGIBILITY:
Group A - Dancers with knee injury:

Inclusion Criteria:

1. Min. 3 hours of classic ballet dancing per week
2. At least 4 years of dancing practice
3. Reported knee pain during the last 6 months

Exclusion Criteria:

1. Injury other than knee joint

Group B - Dancers without knee injury:

Inclusion Criteria:

1. Min. 3 hours of classic ballet dancing per week
2. At least 4 years of dancing practice
3. Reported no musculoskeletal injury during the last 6 months

Exclusion Criteria:

1. None

Group C - Non-dancers athletes:

Inclusion Criteria:

1. Main physical activity is other than dancing

Exclusion Criteria:

1. Reported no musculoskeletal injury during the last 6 months

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: young adolescent female athletes or dancers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Physical evaluation | 1 hour
  Knee range of motion, ligament stability, hypermobility, patella grinding and inhibition test
US - sonographic study of the knee evaluation patellar, tibial and trochlear | 1 hour
  a sonographic study of the knee evaluating patellar, tibial and trochlear cartilage

SECONDARY OUTCOMES:
Visual Analog Score for pain | 1 hour
  VAS score for pain
Function questionnaire | 1 hour
  Questionnaire regarding athletic/dancing activities

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev-Ner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Department of Orthopedic Rehabilitation, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Result] Ivkovic A, Franic M, Bojanic I, Pecina M. Overuse injuries in female athletes. Croat Med J. 2007 Dec;48(6):767-78. doi: 10.3325/cmj.2007.6.767. PMID 18074410
- [Result] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Injury patterns in young, non-professional dancers. J Sports Sci. 2011 Jan;29(1):47-54. doi: 10.1080/02640414.2010.521167. PMID 21086212
- [Result] Tursz A, Crost M. Sports-related injuries in children. A study of their characteristics, frequency, and severity, with comparison to other types of accidental injuries. Am J Sports Med. 1986 Jul-Aug;14(4):294-9. doi: 10.1177/036354658601400409. PMID 3728781
- [Result] Hamilton D, Aronsen P, Loken JH, Berg IM, Skotheim R, Hopper D, Clarke A, Briffa NK. Dance training intensity at 11-14 years is associated with femoral torsion in classical ballet dancers. Br J Sports Med. 2006 Apr;40(4):299-303; discussion 303. doi: 10.1136/bjsm.2005.020941. PMID 16556782
- [Result] Bennell K, Khan KM, Matthews B, De Gruyter M, Cook E, Holzer K, Wark JD. Hip and ankle range of motion and hip muscle strength in young female ballet dancers and controls. Br J Sports Med. 1999 Oct;33(5):340-6. doi: 10.1136/bjsm.33.5.340. PMID 10522638
- [Result] Negus V, Hopper D, Briffa NK. Associations between turnout and lower extremity injuries in classical ballet dancers. J Orthop Sports Phys Ther. 2005 May;35(5):307-18. doi: 10.2519/jospt.2005.35.5.307. PMID 15966542
- [Result] Hamilton WG, Hamilton LH, Marshall P, Molnar M. A profile of the musculoskeletal characteristics of elite professional ballet dancers. Am J Sports Med. 1992 May-Jun;20(3):267-73. doi: 10.1177/036354659202000306. PMID 1636856
- [Result] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Extrinsic and intrinsic risk factors associated with injuries in young dancers aged 8-16 years. J Sports Sci. 2012;30(5):485-95. doi: 10.1080/02640414.2011.647705. Epub 2012 Jan 30. PMID 22288886
- [Result] Coplan JA. Ballet dancer's turnout and its relationship to self-reported injury. J Orthop Sports Phys Ther. 2002 Nov;32(11):579-84. doi: 10.2519/jospt.2002.32.11.579. PMID 12449258
- [Result] Hincapie CA, Morton EJ, Cassidy JD. Musculoskeletal injuries and pain in dancers: a systematic review. Arch Phys Med Rehabil. 2008 Sep;89(9):1819-29. doi: 10.1016/j.apmr.2008.02.020. PMID 18760170
- [Result] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Joint range of motion and patellofemoral pain in dancers. Int J Sports Med. 2012 Jul;33(7):561-6. doi: 10.1055/s-0031-1301330. Epub 2012 May 4. PMID 22562733
- [Result] Witvrouw E, Bellemans J, Lysens R, Danneels L, Cambier D. Intrinsic risk factors for the development of patellar tendinitis in an athletic population. A two-year prospective study. Am J Sports Med. 2001 Mar-Apr;29(2):190-5. doi: 10.1177/03635465010290021201. PMID 11292044
- [Result] Brussaard C, Naudts P, De Schepper A. Ultrasonographic diagnosis of chondromalacia of the femoropatellar joint. J Belge Radiol. 1991;74(4):303-6. PMID 1797798